CLINICAL TRIAL: NCT03739918
Title: Complex Cystic Benign Adrenal Incidentalomas Mimicking Non-adenomatous Masses; Rare Pathologies: Clinical Features and Outcomes. Case Series With Short Review of Literature.
Brief Title: Rare Cystic Benign Adrenal Incidentalomas
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelbaset, principal investigator, Mansoura University
Other Study IDs: adrenal incidentalomas
Record Dates: First submitted 2018-11-08; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Urologic Diseases; Adrenal Tumor
Keywords: Cystic; Adrenal; Incidentaloma; Vascular; Benign
MeSH Terms: conditions — Urologic Diseases; Adrenal Gland Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with adrenal masses: patients with adrenal mass managed by adrenalectomy

SUMMARY:
Benign complex cystic and vascular adrenal tumors comprise a group of lesions characterized by significant rarity. But, their detection is increasing due to improved radiologic imaging techniques. Nevertheless, they are still conflicting with other lesions. the investigators reviewed their experience with complex cystic benign adrenal tumors in adults, review previous reports to determine the appropriate diagnosis and management of these tumors.

DETAILED DESCRIPTION:
Adrenal masses are incidentally found on computed tomography (CT) of the abdomen (so-called "incidentaloma") (AIs) approximately 4% of the time and in 8% in autopsy series. It is important to distinguish benign from malignant. Also, differentiating functioning vs nonfunctioning tumors. The majority of AIs are nonfunctioning , benign lesions account for 82.5% of cases including adenomas (61%), myelolipomas (10%), adrenal cysts (6%), and ganglioneuromas (5.5%), cortisol-secreting adenomas (5.3%), pheochromocytomas (5.1%), adrenocortical carcinomas (4.7%), metastatic lesions (2.5%), and aldosteronomas (1%).

The frequency of adrenal incidentaloma reported in the radiology literature varies according to imaging modality with computed tomography (CT) scans and magnetic resonance imaging (MRI), it ranges from 0.3 to 7%, whereas with ultrasound, it is 0.4-2 %. The evaluation and classification of adrenal vascular tumors and cysts remain a challenging, in spite of, the frequency of detection over the past years has been facilitated by advances in imaging and molecular histopathology. This overlap not only because of their scarcity but because these lesions are often obscured by the extensive hemorrhage. As a result, surgical excision of these lesions has to trend in the last decades.

Because of that, we retrieved our data to determine the clinical features, histopathological pathognomonic features and the long term outcomes for these lesions.

The computerized dedicated database of patients who were treated for adrenal tumors between January 2010 and December 2017 was reviewed. Only patients aged >18 years were included in the study and their files were fully evaluated. The data collected were the age at the time of presentation, clinical features, medical history, adrenal metabolic profile, radiological tumor characteristics, treatment methods, and histopathological characteristics. In all cases, CT with contrast was performed unless contraindicated and MRI was performed. Also, basic hormonal assay including 24-hour urinary cortisol and plasma metanephrines were requested for all cases. Under general anesthesia with fixation of intra-arterial line, patients were explored laparoscopically or via the lumbar incision. Three days postoperative, the patient was discharged unless hormonal replacement therapy is required for a longer period of time. The patients were followed up by metabolic profile and radiologically after 6 and 12 months postoperatively then annually.

ELIGIBILITY:
Inclusion Criteria:

* cases with adrenal tumors above 18 years old with rare histopathology

Exclusion Criteria:

* age less than 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 291 cases diagnosed with adrenal tumors were treated. Demographic criteria of studied cases and different types of pathologies identified . Three cases were diagnosed to have rare cystic and vascular histopathological variant including: cavernous haemangioma, capillary haemangioma and adrenal teratoma.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with rare pathologies and correlation with demographic and radiological data | 7 years
  collection of rare pathologies ,correlation with other review of literature

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt